CLINICAL TRIAL: NCT04576078
Title: Postoperative Analgesic Effect of Orally Administrated Nefopam After a Total Knee Arthroplasty: a Randomized Controlled Trial
Brief Title: Post-operative Analgesic Effect of Oral Nefopam
Acronym: NefPO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 69HCL20_0111; 2020-002955-40 (EudraCT Number)
Record Dates: First submitted 2020-09-29; First posted 2020-10-06 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Postoperative Pain After a Total Knee Arthroplasty
Keywords: Nefopam; Oral; postoperative pain; hyperalgesia; cerebrospinal fluid and plasma concentration; total knee arthroplasty
MeSH Terms: conditions — Pain, Postoperative; Hyperalgesia | interventions — Nefopam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Nefopam has a distinct bitter taste. A taste masking compound non interfering with chemical properties of the drug is used in both arms. Orally given mixture (nefopam or placebo) is prepared by an independent nurse in a separate location and given to a patient in patient's ward.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NEFOPAM 60mg PO/ 8 hours (Experimental): Oral administration of nefopam 60mg 2 hours before the surgery following by 60mg each 8h for 24h.
  Interventions: Drug: Oral nefopam
- Placebo (Placebo Comparator): Oral administration of a placebo 2 hours before the surgery following by one administration each 8h for 24h.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral nefopam — Oral administration of nefopam 60mg 2 hours before the surgery following by 60mg each 8h for 24h. Oral nefopam is prepared ex-tempore from the intravenous formulation adding a taste masking compound by a non-caring nurse following detailed instructions.
  Arms: NEFOPAM 60mg PO/ 8 hours
Drug: Placebo — Oral administration of a placebo 2 hours before the surgery following by one administration each 8h for 24h. Oral placebo is prepared ex-tempore with a taste masking compound by a non-charge nurse following detailed instructions
  Arms: Placebo

SUMMARY:
Primary knee arthroplasty by total prosthesis is a painful surgery, performed on patients with advanced gonarthrosis (stage III), thus already presenting hyperalgesia and hyperalgesia and allodynia. This terrain makes the risk of postoperative hyperalgesia but also of persistent postoperative risk of persistent post-surgical pain.

Nefopam is a non-opioid centrally acting analgesic drug used as a part of multimodal analgesia. The opioid-sparing effect of nefopam is still controversial across various surgical procedures. In France nefopam is only available as a parenteral formulation; however it is often administered orally. There is currently no study addressing the efficacy of oral nefopam for the postoperative pain management including pain prevention.

The investigators conduct a prospective, double-blinded randomized controlled study with the main objective to examine the effect of perioperative orally administered nefopam on postoperative pain after a total knee arthroplasty. Secondary objectives include the quantification of wound allodynia, analysis of adverse events, clinical outcomes, and a pharmacokinetic study of orally given nefopam (plasma and cerebrospinal fluid dosage).

ELIGIBILITY:
Inclusion Criteria:

* adult patients scheduled for a total knee arthroplasty under spinal anesthesia at the Hopital de la Croix Rousse, Hospice Civils de Lyon, France.
* ASA (American Society of Anesthesiology) class between 1 et 3.
* written informed consent

Exclusion Criteria:

* any contraindication for nefopam (known hypersensitivity, past medical history of seizures, urinary retention, benign prostate hyperplasia, angle glaucoma, ischemic cardiomyopathy waiting for revascularization, atrial fibrillation)
* medical conditions known to influence the pharmacokinetics of nefopam (chronic kidney failure with Glomerular Filtration Rate (GFR) <30mL/min/1,73m2, liver failure, current treatment with rifampicin, carbamazepine, azoles fungicides, macrolides)
* current treatment with benzodiazepines, anxiolytics, antidepressants, histamine H1 antagonists, neuroleptics, baclofen, thalidomide, barbiturates
* medical history of gastric or esophageal surgery.
* phenylketonuria
* pregnancy or breastfeeding
* past use of oral nefopam

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-06-29 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Total morphine consumption within 24h after the surgery. | 24 hours after the surgery.
  Total dose of morphine consumed in 24h frame by a patient (PCA and/or additional morphine administration - parenteral or oral)

SECONDARY OUTCOMES:
Hyperalgesia - Pressure Pain Threshold | 24 hours after the surgery
  The pressure pain threshold is determined using a Von Frey monofilaments on both (operated and contralateral) knees 24 hours after incision.
Hyperalgesia - Punctate Pain Intensity | 24 hours after the surgery
  The Punctuate pain intensity is determined using a Von Frey monofilament n°5,88 (60 g/mm2) and a pain scale (0 = no pain, 10 = the worst pain), on both the operated knee and the contralateral knee 24 hours after incision.
Hyperalgesia - Allodynia zone | 24 hours after the surgery
  The extension of allodynia around the wound is measured using a calibrated brush (100 mNewton) 24 hours after incision.
Pain intensity | 24 hours after the surgery and 3 months after the surgery
  Self-reported pain intensity at rest and while moving the operated leg. Each item is scored on a scale ranging from 0 to 10 (0 = no pain, 10 = the worst pain)
Self reported safety outcomes | 24 hours after the surgery
  Nausea and vomiting, unusual sweating, drowsiness, hallucinations, nightmares, palpitations, irritability
Measures Safety outcomes | 24 hours after the surgery
  The incidence of acute urinary retention, and mean cardiac frequency (calculated from the recorded cardiac frequency 3 times a day) are recorded, confusion, acute angle glaucoma.
Pharmacokinetics:Plasmatic and cerebrospinal fluid concentration of nefopam | 2 hours after the first oral administration of nefopam or Placebo.
  Plasmatic and cerebrospinal fluid concentration of nefopam is measured.
Pharmacokinetics:Plasmatic and cerebrospinal fluid concentration of nefopam-beta-D-glucuronide | 2 hours after the first oral administration of nefopam or Placebo.
  Plasmatic and cerebrospinal fluid concentration of nefopam-beta-D-glucuronide is measured.
Pharmacokinetics:Plasmatic and cerebrospinal fluid concentration of nefopam-N-oxyde | 2 hours after the first oral administration of nefopam or Placebo.
  Plasmatic and cerebrospinal fluid concentration of nefopam-N-oxyde is measured.
Pharmacokinetics:Plasmatic and cerebrospinal fluid concentration of nefopam-N-demethyl | 2 hours after the first oral administration of nefopam or Placebo.
  Plasmatic and cerebrospinal fluid concentration of nefopam-N-demethyl is measured.
Pharmacokinetics:Plasmatic and cerebrospinal fluid concentration of Nefopam hydrochloride | 2 hours after the first oral administration of nefopam or Placebo.
  Plasmatic and cerebrospinal fluid concentration of Nefopam hydrochloride is measured.
Persistent postoperative pain - DN4 (or DN2 by phone) | 3 months after the surgery
  The DN4 questionnaire (or DN2 questionnaire if the visit is realized by phone) ("Douleurs Neuropathiques 4/2" = Neuropathic pain 4/2 in french) is recorded to investigate persistent postoperative pain defined as pain on the operated knee 3 months after the surgery.
Persistent postoperative pain - DN4 | 4 months after the surgery
  The DN2 questionnaire ("Douleurs Neuropathiques 2" = Neuropathic pain 2 in french, abbreviated DN4 questionnaire) is recorded by phone if the 3 months visit is realized out of time. If the score is positive (>=3), the DN4 is recorded at hospital within 2 weeks post the 3 months visit.

CONTACTS AND LOCATIONS:
Overall Officials: Frederic AUBRUN, MD/PHD, Principal Investigator — Département d'Anesthésie Réanimation, Hopital de la Croix Rousse
Locations (1):
- Département d'Anesthésie Réanimation, Groupement Hospitalier Nord, Hospices Civils de Lyon, Lyon, France